CLINICAL TRIAL: NCT03350464
Title: Open-label Pilot Study Using Repetitive Transcranial Magnetic Stimulation as a Treatment for Pain in Parkinson's Disease
Brief Title: Repetitive Transcranial Magnetic Stimulation as a Treatment for Pain in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walton Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS024 RG237-18
Record Dates: First submitted 2017-10-20; First posted 2017-11-22 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Neuropathic Pain; Pain
MeSH Terms: conditions — Parkinson Disease; Neuralgia; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain in PD Arm (Experimental): This arm will receive a total 10 sessions of TMS stimulation over 10 weeks. Pre and post intervention scales will be performed on week one and week 10.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive method that uses electromagnetic induction to produce electric currents in the cortex that are strong enough to depolarise neurons sufficiently to trigger action potentials. It is an outpatient based procedure that when used in conjunction with a neuro-navigation system, specific cortical areas can be targeted for greater accuracy and efficacy. In clinical studies, TMS is delivered as trains of pulses (repetitive TMS, rTMS) to prolong its effects. While the exact mechanism of TMS-induced analgesia is unknown, it is thought to regulate the activity of the complex cortical and subcortical networks involved in the processing of painful signals and possibly strengthening the endogenous descending pain modulation system

SUMMARY:
Transcranial magnetic stimulation (TMS) is a procedure that has been shown to improve pain in chronic sufferers. It is a well-tolerated procedure that can be performed on an outpatient basis. It uses a plastic covered coil that sends a magnetic pulse through the skull into the brain and by targeting particular areas in the brain it can be used to help modulate the perception of pain.

The study intends to use this technique to treat such a disabling symptom in patients who suffer from Parkinson's Disease (PD). Initially the aim is to study this technique in ten patients who are suffering from pain and have PD. These patients would initially require an MRI scan which allows us to map the brain and target the correct brain areas for the delivery of the stimulation. The stimulation would be performed over ten sessions and the patients would be assessed by a clinician using well recognized clinical tools.

It is anticipated that there will be a meaningful improvement in pain. It is also anticipated that TMS is a safe technique to use in patients with PD. The study will be used to help plan a future study that compares TMS with sham technique to prove whether TMS could be an option in the treatment of such a disabling condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a diagnosis of Parkinson's Disease.
2. Medical treatment for the movement disorder to be optimized prior to the study.
3. Despite optimum medical therapy neuropathic pain is a major complaint for the patient:

   1. A minimum total score on the King's Pain Scale of 12 or
   2. A minimum subset domain score on Fluctuation-related Pain of 6 or
   3. A minimum subset domain score on Nocturnal pain of 5 or
   4. A minimum subset domain score on Radicular Pain of 3 or
4. No other cause for the pain is identified.
5. Age 18-80
6. Weekly average pain levels of 3/10 or more at the time of entry
7. The patient is capable of and willing to give informed consent for their participation.
8. The patient is capable of and willing to fill in a daily Pain diary during the study.

Exclusion Criteria:

Patients will be excluded from the trial if they:

1. Are suffering from pain not attributable from Parkinson's Disease
2. Are suffering from any neurological or psychiatric disease that could interfere with provision of reliable data (dementia, major depression, drug abuse, alcoholism)
3. Are suffering from a rapidly progressing malignant disease or other systemic disease that is likely to significantly interfere with their participation in the study
4. Are candidates or have been listed for surgery or other major medical intervention requiring hospitalisation and/or rehabilitation (e.g., hip replacement).
5. Have a history of seizures or epilepsy,
6. Require high doses of medication known to lower the threshold for seizures (e.g., amitriptyline > 100mg/d,
7. Have cerebral space occupying lesion,
8. Have a history of severe head injury (associated with a suspicion of brain injury, e.g. resulting in unconsciousness for over 24 hrs)
9. Have metal located in head (e.g. shrapnel, surgical clips, fragments from welding),
10. Have a cochlear implant,
11. Have a cardiac pacemaker in situ,
12. Have a deep brain or vagal nerve stimulator in situ,
13. Are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
No change in the patient's parkinson's disease as measured by Unified Parkinson's Disease Rating Scale III | 10 weeks
  UPDRS III is a clinical scale that measures the severity of the motor symptoms of Parkinson's Disease. No change is expected in the UPDRS III in the patients recruited from the start of the study to the end of the study.

SECONDARY OUTCOMES:
An improvement by a minimum of 30% in the pain caused by Parkinson's Disease as measured by the King's Parkinson's Disease Pain Scale | 10 weeks
  The King's PD Pain Scale measures the patient's pain caused by Parkinson's Disease. An improvement is expected in the pain caused by Parkinson's Disease of at least 30% on the Kings' PD Pain Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, Mersey, United Kingdom

IPD SHARING:
Plan to Share IPD: No